CLINICAL TRIAL: NCT02044783
Title: Identifying and Treating Physical Function Impairment in Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-3021
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity; Physical Impairment
Keywords: Adults; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Behavior Therapy

ARMS (2):
- Behavioral Intervention (Experimental): Behavioral Counseling Intervention: 6 telephone calls that include physical activity goal-setting, tracking,and problem-solving of barriers
  Interventions: Behavioral: Behavioral Counseling
- Usual Care (No Intervention): Monthly mailed print materials on aging topics (that would generally be administered by subjects' primary care clinic). No behavioral counseling.

INTERVENTIONS:
Behavioral: Behavioral Counseling
  Arms: Behavioral Intervention

SUMMARY:
Sedentary older adults are more likely to develop physical function impairments than active older adults. Physical function measured by slow usual gait speed predicts the risk of future falls, disability, institutionalization and mortality. Behavioral physical activity interventions have improved physical activity and physical function, but have not generally been implemented where they may have the most impact -- primary care settings. In part, this is due to the limited time and training for clinical staff to screen for physical function impairment and to treat with physical activity counseling. The proposed scientific goal is to overcome these barriers by adapting an evidence-based screening tool and telephone-based physical activity intervention into primary care settings.

Aim1: Among older adults who screen positive for physical function impairment, to determine the estimated intervention effect size of a 12-week behavioral intervention on physical activity and physical function.

Hypothesis 1a: Physical activity levels will increase more in the intervention vs. usual care group.

Hypothesis 1b: Physical function will increase more in the intervention vs. usual care group.

Aim 2: Among Aim 1 participants and clinical staff who deliver the functional screening and Aim 1 intervention, to evaluate standard implementation science process metrics of reach, acceptability, and implementation

ELIGIBILITY:
Inclusion Criteria:

* Sedentary patients aged 65-85 years who screen positive for physical function impairment (Physical function impairment includes any of the following: time to complete 4-meter walk ≥4.82 seconds (i.e., ≥0.83 meters/second); a reported fall in the past 3 months; or a reported fear of falling)

Exclusion Criteria:

* Inability to walk ≥30 feet without human assistance7
* Dementia, as assessed by either a Folstein Mini-Mental Status Examination <24 or by patient's primary care provider's assessment
* Severe vision loss (legally blind)
* Severe hearing loss
* Medical condition that precludes increasing physical activity per primary care provider's assessment
* Terminal diagnosis per primary care provider's assessment

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Changes in physical activity as determined by accelerometer | 12 weeks
  Subjects' physical activity levels will be determined by accelerometer measures during week 1 and after a 12-week behavioral intervention.
Changes in physical function as assessed by 400-meter walk speed | 12 weeks
  Subjects' physical function will be assessed by 400-meter walk speed before and after 12-week behavioral intervention.
Changes in physical function as assessed by Short Physical Performance Battery | 12 weeks
  Subjects' physical function will be assessed by the Short Physical Performance Battery before and after a 12-week intervention
Change in physical function as assessed by lower extremity strength testing | 12 weeks
  Subjects' physical function will be assessed by lower extremity strength testing before and after a 12-week behavioral intervention .

SECONDARY OUTCOMES:
Evaluation of standard implementation science process of reach | 1 year
  Reach is the percent of patients consented divided by the number eligible.
Assessment of standard implementation science process metrics of acceptability | 1 year
  Acceptability will be assessed through structured surveys.
Assessment of standard implementation science process metrics of implementation | 1 year
  Implementation process will be assessed by structured surveys

CONTACTS AND LOCATIONS:
Overall Officials: Amy Huebschmann, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States